CLINICAL TRIAL: NCT01480869
Title: Randomized Phase III Trial Comparing Conventional Vitamin D Supplementation vs. Vitamin D Supplementation Tailored to Vitamin D Deficiency in Breast Cancer Patients Treated by Neoadjuvant or Adjuvant Chemotherapy.
Brief Title: Study of Vitamin D Supplementation Tailored to Vitamin D Deficiency in Breast Cancer Patients
Acronym: VITACAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITACAL; VA 2010/12 (Other: VA 2010/12); 2010-023459-27 (EudraCT Number)
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Vitamin D supplementation; in neoadjuvant; adjuvant setting
MeSH Terms: conditions — Breast Neoplasms | interventions — Calcium; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional vitamin D and calcium supplementation (Active Comparator): Conventional vitamin D and calcium supplementation with 2 daily OROCAL VITAMINE D3® (500 mg calcium/200 IU cholecalciferol) tablets.
  Interventions: Drug: calcium and cholecalciferol
- vitamin D supplementation tailored to vitamin D deficiency (Experimental): Conventional calcium supplementation with 2 daily OROCAL 500® (500 mg calcium) tablets to suck + vitamin D3 supplementation (UVÉDOSE®, cholecalciferol, 100 000 IU drinkable solution, 2 ml vial) whose schedule of administration depends on vitamin deficiency level:
  * 100 000 IU of vitamin D3 at D1, D15, D28 and D43 if 25OHD level < 10 ng/mL
  * 100 000 IU of vitamin D3 at D1, D15, D28 if 10 ng/mL ≤ 25OHD level < 20 ng/mL
  * 100 000 IU of vitamin D3 at D1 if 20 ng/mL ≤ 25OHD level < 30 ng/mL
  Interventions: Drug: calcium and cholecalciferol

INTERVENTIONS:
Drug: calcium and cholecalciferol — Tablet to suck: calcium 500 mg bid, cholecalciferol 200 IU bid
  Arms: Conventional vitamin D and calcium supplementation
Drug: calcium and cholecalciferol — Tablet: calcium 500 mg bid + 2 ml drinkable solution cholecalciferol 100 000 IU whose schedule of administration depends on vitamin deficiency level:
  * 100 000 IU of vitamin D3 at D1, D15, D28 and D43 if 25-OHD level < 10 ng/mL
  * 100 000 IU of vitamin D3 at D1, D15, D28 if 10 ng/mL ≤ 25-OHD level < 20 ng/mL
  * 100 000 IU of vitamin D3 at D1 if 20 ng/mL ≤ 25-OHD level < 30 ng/mL
  Arms: vitamin D supplementation tailored to vitamin D deficiency

SUMMARY:
The purpose of this study is to compare normalization of vitamin D serum level after 6 months of vitamin D supplementation adjusted to baseline vitamin D serum level vs.conventional vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Breast adenocarcinoma treated by neoadjuvant or adjuvant chemotherapy within 12 months prior to study enrollment
* WHO performance status 0-1
* Age ≥18 years old
* Affiliation to a social security regime or beneficiary of equivalent social protection
* Written informed consent provided before any study specific procedures

Complementary inclusion criterion for randomization

- Proved vitamin D deficiency as defined by serum vitamin D level lower than 30 ng/ml (75 nmol/L).

Exclusion Criteria:

* Metastatic disease
* History or presence of any other malignancy (except curatively treated nonmelanoma skin cancer or in situ cervix carcinoma) ………….

traités dans les 5 ans précédents.

* Contraindication to calcium or cholecalciferol
* Known severe hypersensitivity to vitamin D or to calcium supplementation or to one of the excipients.
* Disease and/or medical conditions accompanied by hypercalcaemia and/or hypercalciuria
* Calcium lithiasis and tissue calcification
* Hypervitaminosis D
* Presence of significant comorbidities:

  i) Uncontrolled endocrine disease ii) Known disorders of calcium phophorus laboratory testing iii) Proved osteopenia or osteoporosis requiring vitamin D and calcium supplements
* Concomitant treatment with other experimental products or another vitamin D calcium treatment
* Pregnancy, breastfeeding or of reproductive potential not using an effective contraceptive method
* Legal inability or restricted legal ability. Medical or psychological conditions not allowing proper study completion or informed consent signature

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the increase in normalization of serum vitamin D level | 6 months
  To compare the increase in normalization of serum vitamin D level adjusted to baseline level in patients receiving either vitamin D supplementation tailored to vitamin D deficiency or conventional vitamin D supplementation.

SECONDARY OUTCOMES:
Baseline vitamin D/calcium status in this patient population | Baseline
Normalization rate of serum 25-OHD level | 12, 18 and 24 months
Normalization rate of serum 25-OHD level in control patients who shift to experimental strategy | 6 months after crossover
Clinical and biological tolerance profile | During treament administration (can last up to 24 months)
  According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.0
Treatment compliance | During treatment administration (can last up to 24 months)
  Treatment compliance will be assessed using a patient record book
Quality of life | 24 months
  Quality of life is assessed using the EORTC QLQ-C30 questionnaire
Impact of study treatments on bone and joint pains induced by aromatase inhibitors | During treatment administration (can last up to 24 months)
Changes in vitamin and calcium biological markers | Up to 24 months
Predictive value of individual biomarkers | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- CRLC Val d'Aurelle-Paul Lamarque, Montpellier, France

REFERENCES:
- [Derived] Jacot W, Firmin N, Roca L, Topart D, Gallet S, Durigova A, Mirr S, Abach L, Pouderoux S, D'Hondt V, Bleuse JP, Lamy PJ, Romieu G. Impact of a tailored oral vitamin D supplementation regimen on serum 25-hydroxyvitamin D levels in early breast cancer patients: a randomized phase III study. Ann Oncol. 2016 Jul;27(7):1235-41. doi: 10.1093/annonc/mdw145. Epub 2016 Mar 30. PMID 27029707